CLINICAL TRIAL: NCT01807884
Title: Comparison of Two Strategies of Oropharyngeal and Tracheal Suctioning in Mechanically Ventilated Patients: a Pilot Trial
Brief Title: Comparison of Two Strategies of Oropharyngeal and Tracheal Suctioning in Mechanically Ventilated Patients
Acronym: AMYLASPI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Teleflex (Industry)
Responsible Party: Principal Investigator, Marion Griton, Doctor Marion Griton, MD, University Hospital, Bordeaux
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: AMYLASPI
Record Dates: First submitted 2013-01-30; First posted 2013-03-08 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Ventilator Acquired Pneumonia; Aspiration
Keywords: Microaspiration; Ventilator acquired Pneumonia; Amylase; Mechanical ventilation; Suction
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimized oral care (Experimental): An optimization of the oropharyngeal suction procedure will include use of a subglottic drainage in a specified order: 1. subglottic suction, 1.oral suction followed by mouth care 3. subglottic suction 4. tracheal suction
  Interventions: Procedure: Optimized oral care
- Routine oral care (Placebo Comparator): Oral suction followed by mouth care and tracheal suction
  Interventions: Other: Routine oral care

INTERVENTIONS:
Procedure: Optimized oral care — An optimization of the oropharyngeal suction procedure will include use of a subglottic drainage in a specified order: 1. subglottic suction, 1.oral suction followed by mouth care 3. subglottic suction 4. tracheal suction
  Arms: Optimized oral care
Other: Routine oral care — Oral suction followed by mouth care and tracheal suction without any subglottic suction
  Arms: Routine oral care

SUMMARY:
The purpose of this study is to evaluate the impact of an optimized suctioning procedure on the risk of endotracheal microaspiration, measured by tracheal to oropharyngeal ratio of amylase enzymatic activity.

DETAILED DESCRIPTION:
• Study design : This is an open prospective, cross-over cohort study, including patients ventilated in one medical intensive care unit. Two procedures will be compared in two distinct, randomly decided cross-over consecutive periods

• Detailed description : Standard cares include tracheal suctions several times a day. They can induce a cough reflex in non paralysed patients leading to the mobilisation of the endotracheal tube and a consecutive raise in the risk of tracheal microaspiration. Thus drainage of subglottic secretion before tracheal suction is expected to reduce microaspiration. Subglottic secretion drainage could decrease the risk of Ventilator Associated Pneumonia even if it remains to be confirmed. However, no study assessed its efficiency in reducing tracheal microaspiration.

An optimization of the oropharyngeal suction procedure will include the use of a subglottic drainage in a specified order to realize a so called "optimized oral care". A comparison will be done with a routine oral care.

We will conduct a crossover study in which the patient's follow-up will last 2 days. Length of suction procedure and mouth care, volume of oral, subglottic and tracheal secretions and their qualitative appearance will be collected. The amylase enzymatic activity will be assessed in oropharyngeal, subglottic and tracheal samples.

• Registry procedure : All requested information will be recorded on case report forms and explanation will be reported for any missing data. False data will be clearly corrected, and signed by investigator or authorised person. For biochemical data (amylase enzymatic activity), results will be transmitted through excel software via a key and data will be integrated to the principal excel file on professional computer of the investigator.

Monitoring will be realised by the co-investigator in association with the clinical research associate.

* Quality factors. This clinical research associates will regularly check data to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry and a report will be report after each checking.
* Sample size assessment: Number of subjects : 24 patients. Six months should be necessary to include these patients.
* Statistical analysis : The sample size estimate assumed a median ratio of 8% and an estimated reduction from 8 to 2% with the optimized oral care. We determined that 12 patients per group would provide a power of 80%, with an α level of 5%.

Results will be expressed as means ± Standard Deviation. Continuous variables will be compared using the Student's t-test for matched paired series and categorical variables using the Chi 2 test. All p values and confidence intervals will be two-tailed. p<0.05 will be considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Intubated with a subglottic secretion drainage device
* ventilated more than 48 hours
* patients yielding a significant tracheal suctioning volume (on a semi-qualitative evaluation: ≥ ++ on a scale consisting of 0,+,++,+++)

Exclusion Criteria:

* paralysed patients
* patients with Ramsay 1, 2
* patients breathing spontaneously
* patients less than 18 years old
* patients in a moribund state
* contra-indication for suctioning procedure (risk of haemorrhage, bronchospasm, Acute Respiratory Distress Syndrome with P/F < 100, malformation or tracheal fistula)
* bronchiectasis, cystic fibrosis, chronic obstructive pulmonary disease
* patients necessitating a closed-suctioning device (prevention of respiratory multiresistant bacteria transmission, Acute Respiratory Distress Syndrome with P/F ratio < 100)
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2016-03-04 (Actual); Study Completion 2016-03-04 (Actual)

PRIMARY OUTCOMES:
tracheal to oropharyngeal ratio of amylase enzymatic activity | Day 1 and Day 2
  As a surrogate for microaspiration, the tracheal to oropharyngeal ratio of amylase enzymatic activity will be assessed after oral care. A mean of measures realized one day after optimized oral care will be compared to a mean of measure realized the other day after standard oral care as a cross over protocol.

SECONDARY OUTCOMES:
volume of the tracheal, subglottic, and oral suctions | three time a day, during 2 days
  qualitative evaluation of volume of the tracheal, oral and when applicable subglottic suctions
length of each mouth care | three time a day, during 2 days
  Length in minutes of each mouth care, including tracheal, oral and when applicable subglottic, suctions
cost of the optimized oral suctioning compared with routine care | At the end of the period of study (48hours) for each patient
  Mean cost of needed material and timed spented by nurses for each mouth care

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Boyer, MD, Principal Investigator — Université Victor Segalen Bordeaux 2
Locations (1):
- Hospital Pellegrin, Bordeaux, Gironde, France

IPD SHARING:
Plan to Share IPD: No